CLINICAL TRIAL: NCT06580886
Title: Validation of Handheld Ultrasound Devices for Point of Care Use in Rheumatology
Brief Title: Validation of Handheld Ultrasound Devices in Rheumatology
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Florida (Other); University Health Network, Toronto (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Sibel Aydin, Professor, Ottawa Hospital Research Institute
Other Study IDs: 20220612-01H
Record Dates: First submitted 2024-08-27; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis; Imaging; Ultrasound
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Psoriatic arthritis: Age ≥18, Meets the classification for psoriatic arthritis (CASPAR) criteria, Able to provide an informed consent, Having peripheral disease phenotype of PsA, At least one tender and swollen join on the day of US
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — All patients having ultrasound with Clarius L15/L20 and GE logic E9/E10 in same visit.

SUMMARY:
The goal of this clinical trial is to test the concurrent validity of the Clarius handheld ultrasound devices versus gold-standard device to detect characteristic features of healthy and rheumatic joints in adults Psoriatic Arthtritis patients (i.e. anatomical structures and vascular flow).

DETAILED DESCRIPTION:
This study is a clinical trial testing the concurrent validity of Clarius handheld ultrasound devices against the gold-standard device to detect characteristics (i.e., anatomical structures and vascular flow) of healthy and rheumatic joints in adult Psoriatic Arthritis patients.

The study will be conducted in 3 centers and 10 patients will be included in each center. Study patients will not be randomized to any group.

Both B mode and Doppler images of the participants' predetermined nail, joint, tendon and enthesitis areas will be recorded with both handheld (Clarius Mobile Health Inc, HD3 L15 scanner, HD3 L20 scanner) and the gold standard device (GE LogicE9/E10) at baseline visit.

Two paper CRFs, patient and physician CRFs, will be filled for each patient during the visit and these will be the source document. The CRFs (eCRFs) will be scanned and uploaded to the SharePoint at each center, within 3 days after the visit. In addition, US images of each patient will be uploaded to the SharePoint. The paper CRFs (source documents) will be kept on site. US images and CRFs uploaded from each center will be reviewed by the research assistant at Ottawa Hospital Research Institute (OHRI) center. If there are any missing or erroneous data in the CRF copy, research assistant will contact the site to ensured that the errors and deficiencies are corrected in source document according to Good Documentation Practice. Site should then re-scan the CRF to the SharePoint, ensuring sequential versioning. Any queries will be confirmed with the site within a week of the data entry. Then the analyzed CRFs data will be transferred to Research Electronic Data Capture (REDCap) ( version 12.4.18 - © 2023 Vanderbilt University) by the research assistant at OHRI. Before each analysis (interim and final), all the paper CRFs and REDCap data will be compared for quality assurance.

The scoring of the US images will be done blindly by the principal investigator at OHRI as stated below.

At the central site (OHRI), the research assistant will give a unique identifier number to each image, for a random quality control and for cross referencing whenever needed. The cropped images, as detailed below, will not have the subject ID visible to the PI at the time of reading but will be accessible for the quality control. (read-only access). The research assistant at OHRI is the only site personnel who has the capacity to uncrop the images in the PowerPoint file (password protected files).

Images will not contain any identifiable information such as Date of Birth (DOB) or initials. The US images will be transferred to a PowerPoint file by the research assistant at OHRI in JPEG format. The research assistant will generate an unblinded master list, inaccessible to other site personnel, to link the slide numbers with the patients and scanned anatomical sites and the slide will have no other information on the patient number or ID. For scoring the images by the PI, a random order slide show will be conducted, irrespective of the machine used or the anatomical site or patient assessed, to ensure blindness to data related to the patient identifiers (The PI will not be blinded to the machine that the image was taken with as the JPEG format that is achieved from different machines are identifiable, but due to the random order scoring, images that belong to the same joint by the different machines are not to be scored consecutively). There will be nine separate powerpoint files, for images of joints, tendons, entheses, nail including power Doppler and gray scale findings; and grey scale file for erosions.

If there are missing images for some sites for any of the probes, the images that were obtained for the same site using other probe(s) will also be excluded. The number of missing joint/tendon/entheses and nail images will be reported. Missing data will not be imputed.

After the images are evaluated blindly, statistical analysis will be completed as described below.

The primary endpoint analysis will be the interrater agreement of detecting any synovitis in B mode with the Clarius and gold standard machine. The kappa coefficients will be evaluated using the guideline outlined by Landis and Koch, where the strength of the kappa coefficients are: 0.01-0.20 slight; 0.21-0.40 fair; 0.41-0.60 moderate; 0.61-0.80 substantial; 0.81-1.00 almost perfect.

For secondary outcomes, the interrater agreement for the presence of Doppler signals within the joints, tenosynovitis, erosions, nail, as well as features of enthesitis (hypoechogenicity, thickening, erosions, enthesophytes, calcifications) will also be evaluated using the same method. The agreement of the semiquantitative grading of the intraarticular findings' severity (synovitis in B mode, Doppler signals, erosions, each being on a scale between 0-3) will be done using weighted kappa analysis.

The study will be completed after the imaging of all patients is completed and the analysis of data is done.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Meets the classification for psoriatic arthritis (CASPAR) criteria
* Able to provide an informed consent
* Having peripheral disease phenotype of PsA
* At least one tender and swollen join on the day of US

Exclusion Criteria:

* Having isolated axial PsA
* Being in MDA with no tender and swollen joints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who fulfilled the inclusion and exclusion criterion.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Intraarticular synovitis scoring | 6 months
  After the imaging of all patients is completed, intraarticular synovitis scoring will be done based on the OMERACT definitions (scales of 0-3) as follows.
  Greyscale inflammatory (hypoechoic) synovial hyperplasia:
  Grade 0: no hypoechoic synovial hyperplasia Grade 1: minimal hypoechoic synovial hyperplasia (filling the angle between the periarticular bones, without bulging over the line linking tops of the bones) Grade 2: hypoechoic synovial hyperplasia bulging over the line linking tops of the periarticular bones but without extension along the bone diaphysis Grade 3: hypoechoic synovial hyperplasia bulging over the line linking tops of the periarticular bones and with extension to at least one of the bone diaphysis

SECONDARY OUTCOMES:
Intraarticular Doppler scoring | 6 months
  After the imaging of all patients is completed, the intraarticular Doppler scoring will be done based on the OMERACT definitions (scales of 0-3).
  Power Doppler signal:
  Grade 0: no flow in the hypoechoic synovial hyperplasia Grade 1: up to three single spots signals or up to two confluent spots or one confluent spot plus up to two single spots Grade 2: vessel signals in less than half of the area of the synovium (≤50%) Grade 3: vessel signals in more than half of the area of the synovium (>50%)
  Also, a lateral view of the 2nd metacarpophalangeal and 5th metatarsophalangeal joints will be recorded in the baseline visit for erosion assessment. Erosions will be described as intra-articular discontinuity of the bony surface seen in 2 perpendicular planes and will be evaluated after the imaging of all patients is completed.
Assessment of nail images | 6 months
  B mode and doppler images of the 2nd nail or most involved nail with all probes (Clarius L20, GE Logic E9/S8) will be recorded in the baseline visit. The loss of the trilaminar appearance and the presence of doppler signal in the nail will be evaluated after the imaging of all patients is completed. During imaging of the nail, if any Doppler signal is detected in nail bed, regardless of its severity, the presence of Doppler signal will be considered positive.
Assessment of tendon images | 6 months
  B mode and Doppler images of the tibialis posterior tendon with Clarius L15 and GE Logic E9/S8 will be recorded in the baseline visit. The presence of tendonitis, tenosynovitis and intratendinous Doppler signal in tibialis posterior tendon will be evaluated after the imaging of all patients is completed.
  B mode and Doppler images of the 2nd extensor digitorum tendon with Clarius L20 and GE Logic E9/S8 will be recorded in the baseline visit. The presence of paratenonitis and intratendinous Doppler signal in the extensor digitorum tendon will be evaluated after the imaging of all patients is completed.
Assessment of entheses images | 6 months
  Elementary lesions of enthesitis will be defined and scored as per the GRAPPA US working group's definitions, as used in the multicenter DUET study.
  All of the elementary lesions will be assessed for their presence or absence. In addition, some of the lesions will also be scored for their severity using a semiquantitative system (grade 0 to 3). The definitions of each grade are outlined below.
  • Hypoechogenicity: Grade 0: Absent Grade 1: Present
  • Thickening: Grade 0: Absent Grade 1: Present
  • Bone Erosion: Grade 0: Absent Grade 1: Present
  • Enthesophyte: Grade 0: No enthesophytes Grade 1: Small enthesophyte Grade 2: Medium enthesophyte Grade 3: Large enthesophytes
  • Calcification: Grade 0: No calcifications Grade 1: Punctate hyperechoic area Grade 2: Linear calcification without acoustic shadow Grade 3: Egg-shell calcification with posterior acoustic shadow
  • Doppler Signal: Grade 0: No Doppler signal Grade 1:A single confluent Doppler signal or

OTHER OUTCOMES:
Adverse event | 6 months
  Adverse events will be recorded during scanning.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Z Aydin, Prof, Principal Investigator — Ottawa Hospital Research Institute; Lihi Eder, Prof, Principal Investigator — Women's College Hospital; Gurjit Kaeley, Prof, Principal Investigator — University of Florida
Locations (3):
- University of Florida College of Medicine, Gainesville, Florida, United States
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Women's College Research Institute, Toronto, Ontario

DOCUMENTS (2):
  • Study Protocol (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT06580886/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT06580886/SAP_001.pdf